CLINICAL TRIAL: NCT00279968
Title: Investigating Significant ICD Heart Therapies Registry Study (INSIGHTS ICD Registry)
Brief Title: INSIGHTS ICD Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Other Study IDs: 231
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
Keywords: ICD; Registry; Ventricular tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: ICD

SUMMARY:
The purpose of the Registry is to collect data on how Implantable Cardioverter Defibrillator (ICD) therapies and medications are being used by physicians to treat ventricular arrhythmias in order to better understand how to improve the clinical care of patients and effectiveness of ICD therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients or legal guardians who are willing and able to sign a Permission for Access to and Use of Health Information in a Registry Form and, if required by an Institution's IRB, an Informed Consent.
* New or replacement implants of Medtronic market released single, dual or triple chamber ICDs including: GEM VR, GEM DR, GEM III AT, Marquis VR, Marquis DR, Maximo DR, Maximo VR, InSync ICD, InSync Marquis ICD and InSync II Marquis ICD.

Exclusion Criteria:

* Patients enrolled in a device study which effects programming and or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1326
Dates: Start 2004-02; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Buxton, MD, Principal Investigator — Rhode Island Hospital
Locations (44):
- United States (44):
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Poway, California
  - Sacramento, California
  - Santa Ana, California
  - Boulder, Colorado
  - Bradenton, Florida
  - Lakeland, Florida
  - Lauderdale Lakes, Florida
  - Palm Beach Gardens, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Chicago, Illinois
  - Crown Point, Indiana
  - Noblesville, Indiana
  - Monroe, Louisiana
  - Annapolis, Maryland
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Columbia, Missouri
  - Omaha, Nebraska
  - Newark, New Jersey
  - Pomona, New Jersey
  - Brooklyn, New York
  - Mineola, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Minot, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Lancaster, Pennsylvania
  - Langhorne, Pennsylvania
  - Providence, Rhode Island
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Fredericksburg, Virginia